CLINICAL TRIAL: NCT04771624
Title: May Covid-19 Impair Executive Functions? A Crossectional Study
Brief Title: Assessment of Executive Functions After Covid-19
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Diyaddin Güleken, Medical Doctor, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: 21022021
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Covid19; Cognitive Impairment
MeSH Terms: conditions — COVID-19; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Subjects who have been Covid positive by RT-PCR at least 60 days ago and not having any symptoms of Covid-19 at the moment
- Healthy: Subjects who do not have any general medical, neurological or psychiatric disorder

SUMMARY:
As it is evident that Covid-19 may have some impacts on cognition, the primary aim of this study is to investigate -if any- deficits of attention, working memory and executive functions after Covid-19.

DETAILED DESCRIPTION:
Since Covid-19 (Coronavirus Disease-2019) was declared as a pandemic by the World Health Organization (WHO) on December 31, 2019, it is still widespread and deadly. As an ongoing pandemic, it has led to a panic and then a controlled fear in societies. In many studies, neuropsychological deficits were observed in Covid-19 patients both during the illness and after recovery. A recent study found that impairment in cognitive functions continued after recovery of Covid-19, and it was associated with peripherical inflammatory markers, such as C-Reactive Protein (CRP). CRP, as a peripherical inflammatory marker, has been proven to be inversely related to serum levels of the brain-derived neurotrophic factor (BDNF), an important neurotrophin in the growth and differentiation of neurons. In this study, attention, working memory and executive functions of Covid-19 patients at post-covid period and its relation with the severity of the disease will be investigated.

ELIGIBILITY:
Inclusion Criteria:

Covid-19 patients:

* Diagnosed as Covid-19 by RT-PCR at least 60 days but not more than 90 days ago
* Asymptomatic at the moment
* Not having any other general medical, neurological or psychiatric conditions except Covid-19 at the time of acute infection

Healthy subjects:

* Not having any of Covid-19 symptoms at the testing time point
* Not having any general medical, neurological or psychiatric condition

Exclusion Criteria:

Covid-19 patients:

* Diagnosed as Covid-19 by RT-PCR less than 60 days or more than 90 days ago
* Having any symptom of acute phase of Covid-19
* Having any other general medical, neurlogical or psychiatric contidions

Healthy subjects:

* Having any of Covid-19 symptoms at the testing time point
* Having any general medical, neurological or psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, 50 healthcare personnel diagnosed as Covid-19 by RT-PCR treated at the Department of Infectious Diseases, Gazi Yaşargil Tranining and Research Hospital, Sağlık Bilimleri Üniversitesi, Diyarbakır, have been randomly recorded and followed up for 60 days, and age, sex, education level and professionally matched 50 healthy subjects randomly recruited from the personnel of the same hospital.
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Neuropsychological test scores | Up to 90 days
  Neuropsychological test scores of Covid-19 patients in comparison with healthy control subjects

SECONDARY OUTCOMES:
Severity of the disease | Up to 90 days
  Neuropsychological test score changes according to the disease severity of Covid-19 patients

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet D Güleken, MD, Principal Investigator — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Sağlık Bilimleri Üniversitesi Gazi Yaşargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All the data of the participants is being declared as it will be preserved, in the informed consent at the point of enrollment

REFERENCES:
- [Background] Wilson BA, Betteridge S, Fish J. Neuropsychological consequences of Covid-19. Neuropsychol Rehabil. 2020 Oct;30(9):1625-1628. doi: 10.1080/09602011.2020.1808483. No abstract available. PMID 32869697
- [Background] Zhou H, Lu S, Chen J, Wei N, Wang D, Lyu H, Shi C, Hu S. The landscape of cognitive function in recovered COVID-19 patients. J Psychiatr Res. 2020 Oct;129:98-102. doi: 10.1016/j.jpsychires.2020.06.022. Epub 2020 Jun 30. PMID 32912598
- [Background] Guo Q, Zheng Y, Shi J, Wang J, Li G, Li C, Fromson JA, Xu Y, Liu X, Xu H, Zhang T, Lu Y, Chen X, Hu H, Tang Y, Yang S, Zhou H, Wang X, Chen H, Wang Z, Yang Z. Immediate psychological distress in quarantined patients with COVID-19 and its association with peripheral inflammation: A mixed-method study. Brain Behav Immun. 2020 Aug;88:17-27. doi: 10.1016/j.bbi.2020.05.038. Epub 2020 May 19. PMID 32416290